CLINICAL TRIAL: NCT01048229
Title: Evaluation of the Tolerance and Acceptability of Rasagiline in the Treatment of Early-stage Parkinson's Disease
Acronym: ACTOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment
Sponsor: Qualissima (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTOR protocol
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Early-stage Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline (Experimental)
  Interventions: Drug: Rasagiline
- Pramipexole (Active Comparator): pramipexole three times daily (titrated from 0.375 mg/day to 1.5 mg/day)
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Rasagiline — 1 mg rasagiline once daily (plus placebo twice daily)
  Arms: Rasagiline
Drug: Pramipexole — pramipexole three times daily (titrated from 0.375 mg/day to 1.5 mg/day)
  Arms: Pramipexole

SUMMARY:
Title: Evaluation of the tolerance and acceptability of Rasagiline in the treatment of early-stage Parkinson's disease.

Type of study: Phase IV

Study objectives:

Principal objective:

To evaluate the tolerance and acceptability of Rasagiline versus Pramipexole (dopamine agonist).

Secondary objectives: To evaluate the clinical benefits of Rasagiline administered as a monotherapy in patients presenting with early-stage Parkinson's disease.

Study design:

Multicentre comparative randomised parallel-group double-blind study, with a total duration of fifteen weeks (three weeks of dose titration and twelve weeks of follow-up), comprising four evaluations (D0, W3, W9, W15).

Number of patients:

240 patients (i.e. 120 in each group) presenting with early stage idiopathic Parkinson's disease.

Number of centres:

70 neurologists distributed throughout three French regions

Treatment studied: Rasagiline Presentation: 1 mg tablets Dosage : 1 mg/day in a single dose, in the morning at breakfast-time.

Comparator: Pramipexole Presentation: 0.125 mg, 0.25 mg and 1 mg pramipexole dihydrochloride monohydrate tablets (corresponding respectively to 0.088 mg, 0.18 mg and 0.7 mg of pramipexole)

Dose-titration: As specified in the SPC for pramipexole, the product will be administered in three daily doses, preferably with meals, and the treatment will begin with a dose-titration phase of three weeks' duration, during which time the dosage will be gradually increased.

On completion of the dose-titration phase, the minimum therapeutic dose of 1.5 mg per day must be achieved by all the patients. The patients who cannot achieve this dosage will be withdrawn from the study. The reason for stopping dose-titration (and leaving the study) will be detailed in the CRF.

Dosage:

The effective dosage of pramipexole should be adapted to the individual, depending on clinical response and tolerance, in successive stages of 0.75 mg at one-week intervals, without exceeding the maximum dose of 3 mg per day.

Treatment prohibited during the study :

Pethidine, fluoxetine, fluvoxamine, dextromethorphan, or any other MAOI, sympathomimetics (including nasal and oral decongestants containing ephedrine or pseudoephedrine), anti-H2s (cimetidine, ranitidine).

Principal evaluation criterion :

The principal criterion of evaluation is the percentage of patients who have presented with at least one " significant " adverse event during follow-up.

A significant adverse event is defined as :

* a severe adverse event (SAE)
* an adverse event which in the opinion of the investigator requires suspension of the treatment or reduction in dosage
* an adverse event considered as severe or moderate by the patient (AEs of which the intensity has not been evaluated will be considered as moderate to severe)

Secondary evaluation criteria:

* analysis of adverse events in the total population
* analysis of adverse events by degree of severity
* analysis of adverse events in subject over 65
* analysis of adverse events by symptom
* percentage of patients presenting with sleep problems (daytime drowsiness, narcolepsy, insomnia, fragmented sleep…)
* evaluation of Epworth Sleepiness Scale
* evaluation of quality of life (PDQ-8)
* evaluation of utilities by EuroQol (EQ-5D)
* overall clinical impression evaluated by the doctor (CGI-I) and by the patient (PGI-I)
* Global-Benefit-Risk (GBR)
* Evaluation of resources

Analysis of the principal criterion:

Analysis of the principal criterion will be carried out with those patients from the intention-to-treat population for whom tolerance data is available in at least one visit after D0.

Comparative analysis The percentages of patients in the two treated groups who present with at least one significant adverse event will be compared using a Khi-2 test.

Logistic regression A logistic regression analysis will be performed in order to explain the presence/absence of a significant event. The nature of the treatment and the centre will act as explanatory variables, and the initial scores as covariates. Analyses will also be performed on quantitative variables (ANCOVA)

Evaluation of the Global Benefit-Risk (GBR) according to the model suggested by Chuang-Stein et al.

Number of subject required:

Calculation of the size is based on the hypothesis that the percentage of patients presenting with at least one significant adverse event during follow-up (principal evaluation criterion) will differ by 15% from one group to the other. With an alpha risk set at 5% and a beta ris kat 20%, the number of subjects required, calculated using the Casagrande et Pike formula, is 110 subjects per group.

The NSN was slightly overestimated in order to maintain the desired strength while taking into account the possibility of lost to follow-up, and was fixed at 240 patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged between 18 and 70
* capable of reading and understanding the information leaflet given to him/her
* signed an inform consent form
* presenting with idiopathic Parkinson's disease with a Hoehn and Yahr score of ≤ 3
* has never been given anti-Parkinson medication, or has been treated with L-Dopa, on condition that the total duration of treatment was less than twelve weeks at a dosage of under 200 mg, or has been treated with a dopamine agonist other than Pramipexole, on condition that:

  * either the patient is still in the dose-titration phase at the time of inclusion
  * or that the treatment was administered for less than six weeks and was completed two weeks before inclusion

Exclusion Criteria:

* women who are pregnant, breastfeeding, or planning a pregnancy in the months after joining the study
* women of reproductive age who have not undergone surgical sterilisation or who are not using a reliable method of contraception before joining the study and during the study
* patient presenting with hepatic insufficiency
* patient presenting with a concommitant illness which is considered significant by the investigator, after examination of the history, the patient's clinical condition, or on the basis on any additional examinations performed
* patient presenting with a skin lesion considered to be suspect by the investigator and which has not been evaluated by a dermatologist
* patient presenting with a contraindication to treatment with Rasagiline or Pramipexole (please see the SPC for the respective products)
* patient treated with fuoxetine during the five weeks preceding inclusion
* patient treated with fluvoxamine, pethidine, selegiline or any other MAOI during the two weeks preceding inclusion
* patient who has had deep brain stimulation treatment
* patient who might receive dextromethorphan or a sympathomimetic during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
frequency of 'significant' adverse events | each visit
  the frequency of 'significant' adverse events up to week 15, defined as a serious adverse event, an adverse event requiring withdrawal of treatment (in the opinion of the investigator) or an event considered as serious by the patient.

SECONDARY OUTCOMES:
percentage of patients with sleep disorders | each visit
  percentage of patients with sleep disorders
Epworth Sleepiness Scale (ESS) | each visit
  Epworth Sleepiness Scale (ESS)
CGI-I and PGI-I | each visit
  Clinical Global Impression of Improvement (CGI-I) scale and the Patient Global Impression of Improvement (PGI-I)